CLINICAL TRIAL: NCT05836376
Title: Is Mitral Annuloplasty an Effective Treatment for Severe Atrial Functional MR?
Status: Completed | Type: Observational
Sponsor: Michele De Bonis (Other)
Responsible Party: Sponsor-Investigator, Michele De Bonis, Chief of Cardiac Surgery of Advanced and Research Therapies, Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Other Study IDs: MAT-SAFMR
Record Dates: First submitted 2023-01-27; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Function Atrial MR
  Interventions: Procedure: Mitral valve annuloplasty
- Functiona Non-atrial MR
  Interventions: Procedure: Mitral valve annuloplasty

INTERVENTIONS:
Procedure: Mitral valve annuloplasty — implantation of a prosthetic ring to treat mitral valve regurgitation

SUMMARY:
Atrial functional mitral regurgitation (MR) is caused by annular dilatation and flattering associated with altered atria/annulus dynamics in patients with severely dilated left atrium and normal leaflets anatomy. Inadequate leaflets adaption is considered a mechanistic culprit as well. Prevalence of at least moderate atrial functional MR varies between 4.7% and 7% in patients with permanent and long standing persistent atrial fibrillation (AF) and is even higher in patients with Heart Failure with preserved Ejection Fraction (HFpEF). Unlike secondary MR in the setting of left ventricular disease, results of surgical treatment of severe atrial functional MR has remained largely unspoken.

The aim of this study is to analyze short and mid-term results of isolated annuloplasty in patients with severe, symptomatic atrial functional MR, in comparission to a matched cohort of patients with secondary MR.

ELIGIBILITY:
Atrial MR group Inclusion criteria

* Adult patients, underwent mitral annuloplasty for atrial functional mitral Anatomical criteria
* Annular dilatation with anterior-posterior diameter (AP) in systole >35mm
* Ratio of AP diameter in systole to anterior leaflet length in diastole >1.3
* Normal leaflets anatomy
* Mild fibrosis may be present
* A small cleft may be present as a result of annular dilatation Functional criteria
* Normal leaflet mobility (Carpentier type I)
* Coaptation depth <10mm
* Absence of ventricular tethering
* Centrality of the regurgitant jet Atrial and ventricular characteristics
* Left atrium diameter > 40 mm
* Normal systolic function of the left ventricle
* Mild left ventricular systolic dysfunction Mild LV (tachycardia induced) with EF >45%
* Absence of regional abnormalities in left ventricular wall motion Clinical criteria
* Persistent, long-standing persistent, or permanent atrial fibrillation

Exclusion criteria

* Degenerative MR including congenital clefts
* LVEF < 45%
* Ventricular tethering
* Coaptation depth >10 mm
* Regional abnormalities in left ventricular wall motion
* Sinus rhythm
* Presence of coronary artery disease
* Absence of annular dilatation

Non-atrial MR group Inclusion criteria

* Adult patients underwent cardiac surgery for non-atrial functional mitral regurgitation in the setting of an idiopathic or ischemic cardiomyopathy

Exclusion criteria

* FE<40%
* Concomitant coronary artery bypass graft
* Age <65 years and >75years
* Treated with annuloplasty + edge-to-edge surgery
* Sinus rhythm

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated for functional mitral regurgitation with annuloplasty. Study group will comprehend patients with atrial functional mitral regurgitation, the control group will be of patients with non-atrial functional mitral regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No